CLINICAL TRIAL: NCT04826562
Title: Switch to DOVATO in Patients Suppressed on Biktarvy (SOUND)
Acronym: Sound
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint Michael's Medical Center (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Jihad Slim, MD, Chief of Infectious Diseases, Saint Michael's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/21
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- dolutegravir/lamivudine (Experimental): dolutegravir/lamivudine
  Interventions: Drug: Dolutegravir/Lamivudine

INTERVENTIONS:
Drug: Dolutegravir/Lamivudine — single tablet antiretroviral
  Other Names: Dovato

SUMMARY:
An open-label, pilot study of switching patients to Dovato who are currently taking Bitarvy who are virological suppressed (HIV-1 < 50 copies/mL

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-1 infection
2. Age of 18 years or older
3. On Biktarvy for at >24 weeks with HIV viral load < 50 copies /mL for > 6 months immediately prior to enrollment
4. Agree to consistently use an effective method of contraception (see Appendix: Highly Effective Methods for Avoiding Pregnancies in Females of Reproductive Potential) for women of child-bearing potential
5. Willingness to sign the informed consent
6. If history of virologic failure must be fully suppressed (HIV-1 RNA<50 copies/mL) for at least 12 months before screening visit
7. No prior HIV genotype or phenotype available

Exclusion Criteria:

1. Hypersensitivity to dolutegravir and/or lamivudine
2. History of virologic failure while on an integrase inhibitor
3. Taking any medication contraindicated for co-administration with dolutegravir and/or lamivudine according to manufacturer's current medication package inserts
4. HIV-1 RNA ≥50 copies/mL (confirmed) in the past 48 weeks after initial suppression on therapy to HIV-1 RNA <50 copies/mL
5. Evidence of Hepatitis B virus (HBV) infection based on the results of testing at screening for Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis B surface antigen antibody (anti-HBs) and HBV DNA as follows:

   * Participants positive for HBsAg are excluded.
   * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.

   Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded. Anti-HBc must be either total anti-HBc or anti-HBc immunoglobulin G (IgG), and NOT anti-HBc IgM. Participants with a documented history of chronic HBV and current undetectable HBV DNA while on a Biktarvy are excluded.
6. Pregnant women, women actively seeking to become pregnant, and women of child-bearing potential who are not using effective contraception
7. Severe hepatic impairment (Child-Pugh C)
8. Critically ill and/or unable to take oral medications
9. Any condition (social or medical) which, in the opinion of the investigator, would make study participation unsafe for the subject
10. Creatinine clearance < 30 mL/min/1.73m2 via CKD-EPI method
11. ALT > 5x the upper limit of normal (ULN) or ALT > 3x ULN and total bilbirubin >1.5x ULN (and >35% directed bilirubin)
12. Subjects with an anticipated need for hepatitis C virus therapy with interferon and/or ribavirin prior to the primary endpoint
13. Unstable liver disease, cirrhosis, and/or known biliary abnormalities (except for hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Virologic Failure | 48 weeks
  To determine the % of virologic failures (VL ≥ 50 copies/mL at week 48 using the FDA ITT, Snapshot analysis

SECONDARY OUTCOMES:
Virologic Suprresion | 96 weeks
  To determine the % of subjects remaining virologically suppressed at weeks 48 and 96 using the Snapshot algorithm
Retrospective Baseline Resistance | 96 weeks
  to determine the percentage baseline resistance after 96 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Michael's Medical Cettner
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No